## Study Survey : Serosurveillance of *B. Pertussis* among children in Kazakhstan

| | PART 1 | _ | |
|---|---|---|---|
| | Date of completion (dd/mm/yyyy): | | |
| | Recruitement Site - Identification Number: | | |
| | Participant - Study Identification Number: | | |
| | QUESTIONS/INSTRUCTIONS | | RESPONSES |
| | Demographics | | |
| 1 | Age of the child | | years |
| 2 | Date of Birth: (dd/mm/yyyy) | | |
| 3 | Sex of the child | | Male<br>Female |
| 4 | Is the child registered in a primary school? | | Yes<br>No |
| | Clinical assessment | | |
| 5 | Have your child had periods of prolonged cough during the last 6 months? | | Yes<br>No |
| 6 | if yes, what is the cough onset date (dd/mm/yyyy if known, otherwise mm/yyyy) | | 11 |
| 7 | if yes (to question 5), have your child had any of these symptom? Whoop post-tussive vomiting Cyanosis | | |
| | Fever | | |
| | Living condition | | 1. In ashaal darmitany |
| 8 | What are the current living arrangements of your child? | | In school dormitory In apartment/house with family Other (Explain) |
| 9 | How many people share the household with your child? | | |
| 10 | Does your child have any roommates? (i.e.do you share a bedroom with anyone) | | Yes<br>No |
| 11 | If yes, how many people share the room? | | NA |
| | | L | |
| | Life style | | |
| 12 | In the last month, were your child exposed to second-hand smoke indoors? | | Yes, every day<br>Yes, some days<br>No, not at all |
| 13 | In the last 6 months, how often have your child visited and stayed in a crowded place (café, mall, kinder nursery | | Never Once per week 2-3 times per week |
| 14 | In the last 6 months, have your child traveled abroad? | | 4 or more times per week Yes No Unknown |
| | Heatlh characterisctics | | |
| 15 | In the past month, have your child taken any antibiotics? (Amoxil, Augmentin, Ciprobay, Zithromax, etc.) | | Yes<br>No<br>Unknown |
| 16 | In the past month, have your child taken any immunosupressants? (i.e.systemic cortisone/prednisone, methotrexate, etc. ) | | Yes<br>No<br>Unknown |

| 17 | In the past month, have your child had any upper respiratory infections? (symptoms of cough, runny nose, or sore throat) | Yes No Unknown |
|---|---|---|
| 18 | Please mark if your child have any of the chronic medical conditions listed? | Diabetes Chronic lung disease* Autoimmune disease* Asplenia (no spleen) Complement deficiency |
| | Vaccination status | |
| 19 | History of vaccination against pertussis | |
| | Date of 1st dose (dd/mm/yyyy): / / Vaccine (brand name): | |
| | Date of 2nd dose (dd/mm/yyyy): / / Vaccine (brand name): | |
| | Date of 3rd dose (dd/mm/yyyy): / / Vaccine (brand name): | |
| 20 | Date of any additional dose (dd/mm/yyyy): / / Vaccine (brand name): | |
| | PART 2: Blood sample and laboratory test | |
| 21 | blood sample initials: | |
| 22 | blood sample taken: | Yes No |
| 23 | Date of blood specimen collection (dd/mm/yyyy): | |
| | Summary of laboratory results | |
| 24 | lg G titer (To Pertussis Toxin) | |
| 25 | lg A titer (To Pertussis Toxin) | |

<sup>\*</sup>Chronic lung disease include: asthma, chronic obstructive pulmonary disease \*Autoimmune disease include: Juvenile arthritis, systemic lupus, Celiac disease